CLINICAL TRIAL: NCT05840978
Title: Effect of Probiotics on Stress in Young Adults: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Probiotics on Stress in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HND-MH-052
Record Dates: First submitted 2023-03-29; First posted 2023-05-03 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Stress
Keywords: Stress; Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotics combined strains (Experimental): Probiotics combined strains administered as oral capsules once daily
  Interventions: Dietary Supplement: Probiotics
- Probiotics single strain (Experimental): Probiotics single strain administered as oral capsules once daily
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Placebo capsule administered orally once daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Oral capsules
  Arms: Probiotics combined strains; Probiotics single strain
Dietary Supplement: Placebo — Oral capsules
  Arms: Placebo

SUMMARY:
The study investigates the effects of probiotics in a young healthy population experiencing stress during a stress challenge, i.e. The Trier Social Stress Test (TSST).

DETAILED DESCRIPTION:
The study is a prospective, randomized, double-blind, three-arm, placebo-controlled study in young adults who are moderately stressed and undergoing a Trier Social Stress Test (TSST), comparing probiotics with placebo. The participants will receive either one of the two test products or placebo daily for a period of eight weeks.

At Visit 1, the participants will be dispensed with study product and complete the Cohen's Perceived Stress Scale (PSS) and State Trait Anxiety Inventory (STAI) questionnaires. Blood samples will be collected for biomarker analysis.

At Visit 2, participants will undergo a TSST and will complete the PSS and STAI questionnaires and Visual Analog Scales (VAS). Saliva and blood samples will be collected for biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed e-consent
* Be between 18 and 45 years old, inclusive
* In general good health, as determined by the investigator
* Have a BMI of ≥18.5 and <30.0 kg/m2
* Willing to consume the study product daily for the duration of the study and comply with the study procedures
* Have moderate stress, as measured on the Cohen's Perceived Stress Scale, with a score between 14 and 26 (inclusive)
* Be able to communicate well with the Investigator, to understand and comply with the study requirements and be judged suitable for the study in the opinion of the investigator

Exclusion Criteria:

* Scores ≥10 on General Anxiety Disorder 7 item (GAD-7) and Patient Health Questionnaire 9 item (PHQ-9)
* Have a history of in-person public speaking or presenting to large groups regularly (≥2 times/year) in the past 12 months
* Have a known major stressful life event occurring (current or upcoming) during the study
* Participants who have a significant illness or condition which may, in the opinion of the investigator impact their ability to participate in the study or impact the study outcomes (e.g. any chronic disease, including hypertension, type 1 or 2 diabetes, cardiovascular diseases, gastrointestinal disorders, celiac disease, and IBD)
* Any disease, that by the investigator's judgement, could interfere with the intestinal barrier function
* Use of oral or systemic (topical allowed) immunosuppressant drugs, antibiotics, steroids, etc. within the one month before screening
* Consumption of probiotic supplements that contain live bacteria in the 4 weeks before the screening
* Regular use of anti-inflammatory drugs such as aspirin or ibuprofen (>200mg/24 hours)
* Food allergy or hypersensitivity to any component of the product
* Heavy alcohol use or recent history (within one year) of illicit drug use
* Participants who work night shifts
* Participation in other clinical trials or studies in the last month
* Desire and/or plans on changing current diet and/or exercise regime during the participation of this study
* Participants who are pregnant or wish to become pregnant during the study
* Participants who are lactating and/or currently breastfeeding
* Participants currently of childbearing potential, but not using an effective method of contraception, as determined by the investigator
* Any Participant who is an employee of the study site or an Atlantia Clinical Trials employee or their close family member or a member of their household

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Perceived stress | Before, during, and after TSST at visit 2 (week 8)
  Change in Perceived Stress Visual Analog Scale (VAS) in response to TSST

SECONDARY OUTCOMES:
STAI score | Before and after TSST at visit 2 (week 8)
  Change in State-Trait Anxiety Index (STAI) in response to TSST. Individual scores on the STAI can range from 40 to 160 with higher scores indicating higher anxiety.
PSS score | baseline and week 8
  Change in Cohen's Perceived Stress Scale (PSS) from baseline to week 8. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
STAI score | baseline and week 8
  Change in State-Trait Anxiety Index (STAI) from baseline to week 8. Individual scores on the STAI can range from 40 to 160 with higher scores indicating higher anxiety.
Anxiety | Before, during, and after TSST at visit 2 (week 8)
  Change in Anxiety Visual Analog Scale (VAS) in response to TSST
Emotional insecurity | Before, during, and after TSST at visit 2 (week 8)
  Change in Emotional Insecurity Visual Analog Scale (VAS) in response to TSST
Exhaustion | Before, during, and after TSST at visit 2 (week 8)
  Change in Exhaustion Visual Analog Scale (VAS) in response to TSST

OTHER OUTCOMES:
Cortisol | Before, during, and after TSST at visit 2 (week 8)
  Salivary cortisol levels in response to TSST
Inflammatory biomarker IL-6 | baseline and week 8
  Blood inflammatory biomarkers from baseline to week 8
Inflammatory biomarker IL-10 | baseline and week 8
  Blood inflammatory biomarkers from baseline to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Professor, Principal Investigator — Atlantia Clinical Trials Ltd
Locations (1):
- Atlantia clinical trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No